CLINICAL TRIAL: NCT04384614
Title: Covid-19 In Tunisia: An Observational Cross-Sectional Registry Study Multicentric Study
Brief Title: Covid-19 In Tunisia: An Observational Cross-Sectional Registry Study
Acronym: CONNAITRE
Status: Withdrawn | Type: Observational
Why Stopped: The sponsor decided to withdraw the study for funding reasons.
Sponsor: Direction des Soins de Santé de Base (Other Government)
Collaborators: Eshmoun Clinical Research Center (Network); Dacima Consulting (Other)
Responsible Party: Principal Investigator, Agnès Hamzaoui, Head of department, Abderrahmane Mami Hospital
Other Study IDs: ECC2020-07
Record Dates: First submitted 2020-05-09; First posted 2020-05-12 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-05

CONDITIONS: Covid 19; BCG Vaccination
Keywords: covid 19; BCG Vaccination
MeSH Terms: conditions — COVID-19 | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — * DNA Check
  * TDR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID (+): Patients COVID19(+) confirmed by PCR
  Interventions: Diagnostic Test: Test PCR; Genetic: TDR; Other: Clinical Examination
- COVID (-): Patients COVID19 (-) who had been in contact with COVID-19 (+) confirmed by PCR
  Interventions: Diagnostic Test: Test PCR; Genetic: TDR; Other: Clinical Examination

INTERVENTIONS:
Diagnostic Test: Test PCR — Viral load (COVID+) testing by PCR
Genetic: TDR — IDR and blood sampling for testing DNA Cheque
Other: Clinical Examination — COVID 19 symptoms and Physical Examination

SUMMARY:
Covid-19 In Tunisia: AN Observational Cross-Sectional Registry Study

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 (+), inpatient or outpatient, confirmed by PCR test
* COVID-19 (-) confirmed by PCR test having been in contact with COVID-19 (+)

Exclusion Criteria:

* COVID(+) and COVID(-) diagnosed by other tests than PCR
* COVID-19 (-) Not having been in contact with COVID19(+)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 Patients will be included between COVID19 (+) and COVID19 (-) patients who have been in contact with COVID19 (+)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Differences related to epidemiological demographic characteristics | 30 days
  Identify differences related to epidemiological demographic characteristics and the profile of COVID(+) vs. the profile of COVID(-) patients who have been in contact with COVID(+)
  * Vaccination History Questionnaire
  * Medical and Surgical History Questionnaire
  * Clinical Examination
  * TDR and blood sampling for DNA Checks

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Hamzaoui, Pr, Principal Investigator — Hopital Abderrahmane Mami
Locations (1):
- Eshmoun Clinical Research Centre, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No